CLINICAL TRIAL: NCT02221466
Title: Measurements of Endothelial Function by Means of Peripheral Arterial Tonometry in Diabetic Foot Ulcer Patients Undergoing Hyperbaric Oxygen Therapy.
Brief Title: Measurement of Endothelial Function With Peripheral Arterial Tonometry in Patients Undergoing Hyperbaric Oxygen Therapy
Status: Completed | Type: Observational
Sponsor: Ole Hyldegaard (Other)
Responsible Party: Sponsor-Investigator, Ole Hyldegaard, Associate Professor, Medical Director, MD, Ph.D, DMSci, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: ENDOPAT-1-HBO-MH-2014
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Diabetic Peripheral Vascular Disease
Keywords: diabetes; foot; wounds; nitric oxide; endothelium; infection; biological markers; observational study; hyperbaric oxygen; ulcers; cytokines; inflammation
MeSH Terms: conditions — Diabetes Mellitus; Wounds and Injuries; Infections; Ulcer; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- diabetic patients: Diabetic patients given HBOT
- None diabetic patients: None diabetic patients given HBOT

SUMMARY:
The purpose of this clinical study is to test whether or not patients treated with HBOT for diabetic foot ulcers will demonstrate measurable changes of the blood vessel function during the course of HBOT treatments. , i.e. an expected increase in the reactive hyperemic index (RHI) measured by the peripheral arterial tonometry (PAT).

DETAILED DESCRIPTION:
Measurement and monitoring of endothelial function can be used for prediction of outcome in acute, severe disease. Diabetic patients have a poorer peripheral vascular function measured by peripheral arterial tonometry (PAT) as compared to normals, but the effect of hyperbaric oxygen therapy (HBOT) on endothelial function in these patients is unknown. Measurement of PAT in patients with diabetic foot ulcers undergoing HBOT, may help to improve treatment and changes in the reactive hyperemic index (RHI) might correlate with wound healing in these patients.

Peripheral arterial tonometer (PAT) has been shown to be an easy, fast and standardized method for measuring the peripheral arterial endothelial function. The method is also operator-independent and has a high reproducibility.

The PAT apparatus (ENDOPAT) measures the post-ischemic response to a five-minute blood flow occlusion of the upper arm, and the relationship between the pre-and post-ischemic pulse amplitude is expressed as a reactive hyperemic index (RHI). The normal RHI in young healthy persons is more than 2, while in critically ill patients and patients with diabetes, hypertension or heart disease it is significantly decreased.

The study aims to test whether or not patients treated with HBOT for diabetic foot ulcers will demonstrate an improvement of the endothelial function in the peripheral vessels, i.e. an increase in RHI measured by the PAT. Similarly, essential mediators of angiogenesis and nitric oxide bioavailability will be measured in peripheral blood taken during the PAT measurements which will be performed at the time of inclusion, before HBOT and subsequently for each 10th HBOT session.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with foot ulcer
* None diabetic patients
* Age > 18 years
* Patients referred to hyperbaric oxygen therapy.
* Patients who have given written informed consent to participate in the study

Exclusion Criteria:

* Patients who cannot cooperate to participate in the study
* Patients who do not understand or speak Danish or English
* Allergy to the materials used in the experiment.
* Patients < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic and none diabetic patients admitted for HBOT.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01-21 (Actual); Study Completion 2016-01-21 (Actual)

PRIMARY OUTCOMES:
Peripheral arterial tonometry (PAT) | 6 weeks
  Changes in PAT measurements upon completion of HBOT sessions.
Peripheral arterial tonometry (PAT) | 18 weeks
  Changes in PAT measurements upon completion of HBOT sessions after 12 weeks.

SECONDARY OUTCOMES:
Nitric oxide and cytokine expression | 6 weeks
  Measurement of nitric oxide bioavailability and levels of cytokine expression levels in serum after HBOT completion.
Nitric oxide and cytokine expression | 18 weeks
  Measurement of nitric oxide bioavailability and levels of cytokine expression levels in serum after HBOT completion following 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Hyldegaard, MD, DMSci, Principal Investigator — University Hospital Copenhagen, Rigshospitalet
Locations (1):
- University Hospital of Copenhagen - Rigshospitalet, Copenhagen, Capitol Region, Denmark

REFERENCES:
- [Background] Londahl M, Katzman P, Nilsson A, Hammarlund C. Hyperbaric oxygen therapy facilitates healing of chronic foot ulcers in patients with diabetes. Diabetes Care. 2010 May;33(5):998-1003. doi: 10.2337/dc09-1754. PMID 20427683
- [Background] Patvardhan EA, Heffernan KS, Ruan JM, Soffler MI, Karas RH, Kuvin JT. Assessment of vascular endothelial function with peripheral arterial tonometry: information at your fingertips? Cardiol Rev. 2010 Jan-Feb;18(1):20-8. doi: 10.1097/CRD.0b013e3181c46a15. PMID 20010335
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Brant LC, Barreto SM, Passos VM, Ribeiro AL. Reproducibility of peripheral arterial tonometry for the assessment of endothelial function in adults. J Hypertens. 2013 Oct;31(10):1984-90. doi: 10.1097/HJH.0b013e328362d913. PMID 23751970
- [Background] Bergstrom A, Staalso JM, Romner B, Olsen NV. Impaired endothelial function after aneurysmal subarachnoid haemorrhage correlates with arginine:asymmetric dimethylarginine ratio. Br J Anaesth. 2014 Feb;112(2):311-8. doi: 10.1093/bja/aet331. Epub 2013 Oct 1. PMID 24085770
- [Background] Mahmud FH, Van Uum S, Kanji N, Thiessen-Philbrook H, Clarson CL. Impaired endothelial function in adolescents with type 1 diabetes mellitus. J Pediatr. 2008 Apr;152(4):557-62. doi: 10.1016/j.jpeds.2007.08.044. Epub 2007 Nov 5. PMID 18346515
- [Background] Moerland M, Kales AJ, Schrier L, van Dongen MG, Bradnock D, Burggraaf J. Evaluation of the EndoPAT as a Tool to Assess Endothelial Function. Int J Vasc Med. 2012;2012:904141. doi: 10.1155/2012/904141. Epub 2012 Feb 14. PMID 22500237
- [Background] Eisenbud DE. Oxygen in wound healing: nutrient, antibiotic, signaling molecule, and therapeutic agent. Clin Plast Surg. 2012 Jul;39(3):293-310. doi: 10.1016/j.cps.2012.05.001. Epub 2012 Jun 2. PMID 22732377
- [Background] Boykin JV Jr, Baylis C. Hyperbaric oxygen therapy mediates increased nitric oxide production associated with wound healing: a preliminary study. Adv Skin Wound Care. 2007 Jul;20(7):382-8. doi: 10.1097/01.ASW.0000280198.81130.d5. PMID 17620739